CLINICAL TRIAL: NCT05008913
Title: A Phase I, Open-Label, Non-Randomised Study of the Absorption, Distribution, Metabolism, and Excretion of Adavosertib After a Single Oral Dose of [14C]Adavosertib to Patients With Advanced Solid Tumours
Brief Title: Human Absorption, Distribution, Metabolism, and Excretion Study of [14C]Adavosertib
Acronym: ADME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated because the clinical development programme for Adavosertib has been discontinued
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D601HC00004
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumors
Keywords: Absorption; Distribution; Metabolism; Excretion; Pharmacokinetics
MeSH Terms: interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]Adavosertib (Experimental): Patients will receive a single administration of [14C]adavosertib as an oral solution on Day 1.
  Interventions: Drug: [14C]Adavosertib

INTERVENTIONS:
Drug: [14C]Adavosertib — Patients will receive a single administration of [14C]Adavosertib as an oral solution on Day 1.
  Other Names: AZD1775

SUMMARY:
This is a non-randomised study in patients with advanced solid malignancies

DETAILED DESCRIPTION:
The aim is to recruit approximately 8 patients with a minimum number of 4 pharmacokinetics (PK) evaluable patients.

Each patient will be admitted to the study site pre-dose on Day -1 and will remain at the study site until at least Day 8. Patients will receive a single administration of [14C]adavosertib as an oral solution on Day 1. During this study, whole blood, plasma, urine, faeces, and vomit samples (if presented) will be collected at various time points to characterise the absorption, distribution, metabolism, excretion and PK of adavosertib.

The duration of the residential period will be evaluated following treatment of the first patient and may be adjusted to ensure recovery of at least 90% of the total radioactivity following the dose of [14C]adavosertib and/or until less than 1% of dose is recovered in urine and/or faeces within a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 years of age.
2. Histologically or cytologically documented, locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
3. Eastern Cooperative Oncology Group performance status score of 0 to 1.
4. Life expectancy ≥ 12 weeks.
5. Patients must have normal organ and marrow function at baseline, within 7 days prior to study drug administration.
6. Able and willing to stay in hospital for approximately 9 days (first patient; to be evaluated and possibly adjusted for subsequent patients) for the collection of samples following a single oral dose of [14C]-adavosertib.
7. Body weight within 50-100 kg and BMI within the range 18-30 kg/m^2 (inclusive).
8. Regular bowel movements (i.e., on average production of at least 1 faeces per day).
9. Males and females of childbearing potential who agree to use contraceptive measures consistent with local regulations for clinical studies.

Exclusion Criteria:

1. Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade > 2) caused by previous anticancer therapy, excluding alopecia and CTCAE Grade 2 peripheral neuropathy.
2. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of 14C-adavosertib oral solution.
3. Patients who have participated in another absorption, distribution, metabolism and excretion study within 1 year prior to screening.
4. Any significant cardiac diseases currently or within the last 6 months such as:

   1. unstable angina pectoris
   2. acute myocardial infarction, congestive heart failure
   3. conduction abnormality not controlled with pacemaker or medication
   4. significant ventricular or supraventricular arrhythmias
5. Any of the following: History or current evidence of congenital long QT syndrome; concomitant medications known to prolong QT interval or history of medication-related QT prolongation.
6. Known to have tested positive for human immunodeficiency virus or active tuberculosis infection.
7. Known active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening.
8. Any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant, active infections, and active bleeding diseases) which prohibit participating in the study.
9. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study intervention.
10. Use of an anti-cancer treatment drug ≤ 21 days (≤ 6 weeks for nitroureas or mitomycin C) or use of an investigational product within 5 half-lives prior to the first dose of adavosertib.
11. Patient uses drugs that are sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or are moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks or 5 halflives (whichever is longer) prior to Day 1 of dosing.
12. Receipt of live virus and live bacterial vaccines whilst the patient is receiving the study intervention and during the 30-day follow-up period. Inactivated flu vaccines are permitted.
13. Any known hypersensitivity or contraindication to the components of the study intervention adavosertib.
14. Currently pregnant (confirmed with positive pregnancy test) or breast feeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Amount and cumulative amount excreted and expressed as the percentage of the administered dose into the urine and faeces from time t1 to time t2 | Urine and fecal samples collected from pre-dose to 168 hours post-dose
  Assessment of the mass balance of total radioactivity, including the routes and rates of elimination following a single oral dose [14C]adavosertib.
Renal clearance of radioactivity (CLR) | From pre-dose to 168 hours post-dose
  Assessment of renal clearance of adavosertib, including the routes and rates of elimination following a single oral dose [14C]adavosertib.
Maximum observed plasma concentration (Cmax) | From pre-dose to 168 hours post-dose
  Assessment of Cmax of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Area under plasma concentration-time curve from time zero to infinity (AUCinf) | From pre-dose to 168 hours post-dose
  Assessment of AUCinf of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Area under the plasma concentration-time curve from zero to time of last quantifiable concentration (AUClast) | From pre-dose to 168 hours post-dose
  Assessment of AUClast of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Time to reach peak or maximum observed concentration following drug administration (tmax) | From pre-dose to 168 hours post-dose
  Assessment of tmax of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Terminal elimination rate constant (λz) | From pre-dose to 168 hours post-dose
  Assessment of λz of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | From pre-dose to 168 hours post-dose
  Assessment of t½λz of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | From pre-dose to 168 hours post-dose
  Assessment of CL/F of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Mean Residence Time of the unchanged drug in the systemic circulation (MRTinf) | From pre-dose to 168 hours post-dose
  Assessment of MRTinf of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Volume of distribution (apparent) at steady state following extravascular administration (Vss/F) | From pre-dose to 168 hours post-dose
  Assessment of Vss/F of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | From pre-dose to 168 hours post-dose
  Assessment of Vz/F of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.
Ratio of AUCinf of plasma adavosertib relative to AUCinf of plasma total radioactivity [AUCinf Plasma:Total Plasma Ratio] | From pre-dose to 168 hours post-dose
  Assessment of AUCinf plasma adavosertib:Total plasma radioactivity ratio following a single oral dose of [14C]adavosertib.
Ratio of AUCinf of whole blood total radioactivity to AUCinf of plasma total radioactivity [AUCinf Blood:Plasma Ratio] | From pre-dose to 168 hours post-dose
  Assessment of AUCinf Blood:Plasma Ratio total radioactivity following a single oral dose of [14C]adavosertib.
Amount, cumulative amount, and cumulative percentage of unchanged adavosertib excreted into urine from time t1 to time t2 | Urine collected from pre-dose to 168 hours post-dose
  Assessment of unchanged adavosertib following a single oral dose of [14C]adavosertib.
Renal clearance of adavosertib from plasma (CLR) | From pre-dose to 168 hours post-dose
  Assessment of CLR of adavosertib and total radioactivity following a single oral dose of [14C]adavosertib.

SECONDARY OUTCOMES:
Number of patients with adverse events (AE) and serious AEs (SAE) | From screening (Day -28 to Day -1) until end of study (within 30 [±7] days of adavosertib dose)
  Assessment of the safety and tolerability of adavosertib following oral dosing in patients with advanced solid tumours.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home